CLINICAL TRIAL: NCT03964519
Title: Neuromuscular, Physiological and Performance Changes After an Acute and Chronic Training Protocol Associated to the Inter-set Velocity Loss
Brief Title: Effects of an Acute and Chronic Training Protocol Associated to the Inter-set Velocity Loss
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Alejandro Muñoz López (Other)
Responsible Party: Sponsor-Investigator, Alejandro Muñoz López, Associate Professor, University of Seville
Organization: University of Seville (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: TMG_velocity_lost
Record Dates: First submitted 2019-05-23; First posted 2019-05-28 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Healthy
Keywords: velocity loss; Tensiomiography; resistance training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 20% velocity loss (Experimental): This group will train with a variable number of repetitions during each set. The group will stop the set once the mean propulsive velocity will be 20% less compared to the first repetition.
  Interventions: Other: Acute changes; Other: Chronic changes; Other: Familiarization
- 40% velocity loss (Experimental): This group will train with a variable number of repetitions during each set. The group will stop the set once the mean propulsive velocity will be 40% less compared to the first repetition.
  Interventions: Other: Acute changes; Other: Chronic changes; Other: Familiarization
- Control group (Placebo Comparator): This group will be just tested as a control group.
  Interventions: Other: Chronic changes; Other: Familiarization

INTERVENTIONS:
Other: Acute changes — In a crossover design, participants will be randomized to perform on Day 1, 3 sets of repetitions (depending on each treatment group) at 70% or 1RM in the full squat exercise. 48-h later, same will be performed but in the contrary crossover arm.
  Arms: 20% velocity loss; 40% velocity loss
Other: Chronic changes — In a randomized control trial, participants will train during 6 weeks the full squat exercise, 2 days in the week (minimum between-days rest of 48h). Intensity will vary from 70% to 85 of 1RM, and training volume from 3 to 6 sets.
Other: Familiarization — Prior to any intervention, all participants will perform a familiarization of the exercise session, together with a progressive resistance test to estimate the 1 RM

SUMMARY:
This study evaluates different performance, physiological and neuromuscular changes after acute and chronic resistance training intervention in physically active men. The participants will train with a single exercise (full squat) and will be monitored with a linear encoder. The experiment will consist of between 3 to 6 sets between 70% to 85% of 1RM in the full squat exercise. Two main groups will form the intervention: one group will perform inter-set repetitions until there will be a 20% of velocity loss compared to the first repetition, while the second group will have a 40% of velocity loss.

DETAILED DESCRIPTION:
The main dependent variables and instruments will be:

1. Tensyomiography: neuromuscular properties of the vastus lateral (VL), rectus femoris (RF) and vastus medialis (VM) from the dominant leg.
2. Force platform: kinetic variables in relation to a countermovement jump.
3. Near-infrared spectrography: oxygen saturation in the VL and VM.
4. Termographic camera: low limbs temperatura.
5. Linear encoder: mean propulsive velocity from each repetition
6. Electromyography: amplitude and frequency parameters related to a knee extension maximum voluntary contraction test.
7. Strain gauge: maximum isometric force.

ELIGIBILITY:
Inclusion Criteria:

* To be healthy
* Without injuries or actual illnesses
* More than 2 years of experience in resistance training or federative sports

Exclusion Criteria:

* To be sick or injured
* To have programmed during the intervention phase a dramatic change in the lifestyle

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2019-08-30 (Estimated); Study Completion 2019-09-15 (Estimated)

PRIMARY OUTCOMES:
Contraction time | 7 weeks
  Time between 10% to 90% on the displacement-time curve assessed with the Tensiomiograhpy
Maximum displacement | 7 weeks
  Maximum displacement point the displacement-time curve assessed with the Tensiomiograhpy

SECONDARY OUTCOMES:
Kinetic variables in the jump | 7 weeks
  Kinetic variables related to the force-time curve registered with the force platform during jumps
Muscle tissue oxygen | 7 weeks
  Oxygen in the muscle tissue assessed via near-infrared spectroscopy
Muscle temperature | 7 weeks
  Low limb muscles temperature assessed with a termographic camera
Mean propulsive velocity | 7 weeks
  Individual repetitions mean propulsive velocity during the full squat exercise, assessed with a linear encoder
Amplitude (RMS) and frequency outputs | 7 weeks
  Muscle electrical activity assessed with an EMG
Peak isometric force | 7 weeks
  Maximum force achieved during a knee extension at 120º

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Muñoz López, PhD, Study Director — Internship; Jesus Gustavo Ponce, PhD, Principal Investigator — Professor

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pareja-Blanco F, Rodriguez-Rosell D, Sanchez-Medina L, Ribas-Serna J, Lopez-Lopez C, Mora-Custodio R, Yanez-Garcia JM, Gonzalez-Badillo JJ. Acute and delayed response to resistance exercise leading or not leading to muscle failure. Clin Physiol Funct Imaging. 2017 Nov;37(6):630-639. doi: 10.1111/cpf.12348. Epub 2016 Mar 11. PMID 26970332
- [Background] Pareja-Blanco F, Rodriguez-Rosell D, Sanchez-Medina L, Sanchis-Moysi J, Dorado C, Mora-Custodio R, Yanez-Garcia JM, Morales-Alamo D, Perez-Suarez I, Calbet JAL, Gonzalez-Badillo JJ. Effects of velocity loss during resistance training on athletic performance, strength gains and muscle adaptations. Scand J Med Sci Sports. 2017 Jul;27(7):724-735. doi: 10.1111/sms.12678. Epub 2016 Mar 31. PMID 27038416
- [Background] Moran-Navarro R, Martinez-Cava A, Sanchez-Medina L, Mora-Rodriguez R, Gonzalez-Badillo JJ, Pallares JG. Movement Velocity as a Measure of Level of Effort During Resistance Exercise. J Strength Cond Res. 2019 Jun;33(6):1496-1504. doi: 10.1519/JSC.0000000000002017. PMID 29944141
- [Background] Sanchez-Medina L, Pallares JG, Perez CE, Moran-Navarro R, Gonzalez-Badillo JJ. Estimation of Relative Load From Bar Velocity in the Full Back Squat Exercise. Sports Med Int Open. 2017 Mar 28;1(2):E80-E88. doi: 10.1055/s-0043-102933. eCollection 2017 Feb. German. PMID 30539090
- [Background] Gonzalez-Badillo JJ, Yanez-Garcia JM, Mora-Custodio R, Rodriguez-Rosell D. Velocity Loss as a Variable for Monitoring Resistance Exercise. Int J Sports Med. 2017 Mar;38(3):217-225. doi: 10.1055/s-0042-120324. Epub 2017 Feb 13. PMID 28192832
- [Background] Rodriguez-Rosell D, Yanez-Garcia JM, Torres-Torrelo J, Mora-Custodio R, Marques MC, Gonzalez-Badillo JJ. Effort Index as a Novel Variable for Monitoring the Level of Effort During Resistance Exercises. J Strength Cond Res. 2018 Aug;32(8):2139-2153. doi: 10.1519/JSC.0000000000002629. PMID 29781942
- [Background] Franz A, Behringer M, Harmsen JF, Mayer C, Krauspe R, Zilkens C, Schumann M. Ischemic Preconditioning Blunts Muscle Damage Responses Induced by Eccentric Exercise. Med Sci Sports Exerc. 2018 Jan;50(1):109-115. doi: 10.1249/MSS.0000000000001406. PMID 28832392
- [Background] Rusu LD, Cosma GG, Cernaianu SM, Marin MN, Rusu PF, Ciocanescu DP, Neferu FN. Tensiomyography method used for neuromuscular assessment of muscle training. J Neuroeng Rehabil. 2013 Jul 3;10:67. doi: 10.1186/1743-0003-10-67. PMID 23822158
- [Background] Gutierrez-Vargas R, Martin-Rodriguez S, Sanchez-Urena B, Rodriguez-Montero A, Salas-Cabrera J, Gutierrez-Vargas JC, Simunic B, Rojas-Valverde D. Biochemical and Muscle Mechanical Postmarathon Changes in Hot and Humid Conditions. J Strength Cond Res. 2020 Mar;34(3):847-856. doi: 10.1519/JSC.0000000000002746. PMID 30024483
- [Background] Wiewelhove T, Raeder C, de Paula Simola RA, Schneider C, Doweling A, Ferrauti A. Tensiomyographic Markers Are Not Sensitive for Monitoring Muscle Fatigue in Elite Youth Athletes: A Pilot Study. Front Physiol. 2017 Jun 16;8:406. doi: 10.3389/fphys.2017.00406. eCollection 2017. PMID 28670284
- [Background] Piqueras-Sanchiz F, Martin-Rodriguez S, Martinez-Aranda LM, Lopes TR, Raya-Gonzalez J, Garcia-Garcia O, Nakamura FY. Effects of moderate vs. high iso-inertial loads on power, velocity, work and hamstring contractile function after flywheel resistance exercise. PLoS One. 2019 Feb 7;14(2):e0211700. doi: 10.1371/journal.pone.0211700. eCollection 2019. PMID 30730959
- [Background] de Paula Simola RA, Harms N, Raeder C, Kellmann M, Meyer T, Pfeiffer M, Ferrauti A. Assessment of neuromuscular function after different strength training protocols using tensiomyography. J Strength Cond Res. 2015 May;29(5):1339-48. doi: 10.1519/JSC.0000000000000768. PMID 25474337
- [Background] Macgregor LJ, Hunter AM, Orizio C, Fairweather MM, Ditroilo M. Assessment of Skeletal Muscle Contractile Properties by Radial Displacement: The Case for Tensiomyography. Sports Med. 2018 Jul;48(7):1607-1620. doi: 10.1007/s40279-018-0912-6. PMID 29605838
- [Background] Raeder C, Wiewelhove T, Simola RA, Kellmann M, Meyer T, Pfeiffer M, Ferrauti A. Assessment of Fatigue and Recovery in Male and Female Athletes After 6 Days of Intensified Strength Training. J Strength Cond Res. 2016 Dec;30(12):3412-3427. doi: 10.1519/JSC.0000000000001427. PMID 27093538
- [Background] Giovanelli N, Taboga P, Rejc E, Simunic B, Antonutto G, Lazzer S. Effects of an Uphill Marathon on Running Mechanics and Lower-Limb Muscle Fatigue. Int J Sports Physiol Perform. 2016 May;11(4):522-9. doi: 10.1123/ijspp.2014-0602. Epub 2015 Sep 21. PMID 26390075